CLINICAL TRIAL: NCT01400737
Title: Oral Ibuprofen Prophylaxis for Patent Ductus Arterioses in Very Extremely Low Birth Weight Infants
Acronym: OIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: H. Gozde Kanmaz, MD, Fellow of Neonatology, Zekai Tahir Burak Maternity Teaching Hospital, Neonatal Intensive Care Unit
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2011-09-ibuprofen; 2011-09 (Other: Zekai Tahir Burak Maternity Teaching Hospital)
Record Dates: First submitted 2011-07-19; First posted 2011-07-22 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Oral Ibuprofen Prophylaxis in Very Low Birth Weight Infants
Keywords: ibuprofen; prophylaxis; VELBW
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- ibuprofen (Experimental): The patients in the control group were given 3 doses of an orange starch suspension as placebo that looked like ibuprofen.
  Interventions: Drug: ibuprofen

INTERVENTIONS:
Drug: ibuprofen — The prophylaxis group received ibuprofen suspension at a dosage of 10 mg/kg via an orogastric tube, followed by 0.5 ml of distilled water. The first dose was given within the first 24 hours of life. The second and third doses were given within 24 and 48 hours after the first dose respectively.
Drug: ibuprofen — The prophylaxis group received ibuprofen suspension at a dosage of 10 mg/kg via an orogastric tube, followed by 0.5 ml of distilled water. The first dose was given within the first 24 hours of life. The second and third doses were given within 24 and 48 hours after the first dose respectively

SUMMARY:
Patent ductus arterioses (PDA) is a major morbidity in preterm infants, especially in extremely premature infants less than 28 weeks. The clinical signs and symptoms of PDA in preterm infants are non specific and insensitive for making an early diagnosis of significant ductal shunting. Functional echocardiography is emerging as a new valuable bedside tool for early diagnosis of hemodynamically significant ductus, even though there are no universally accepted criteria for grading the hemodynamic significance. Echocardiography has also been used for early targeted treatment of ductus arterioses, though the long term benefits of such strategy are debatable. The biomarkers like BNP and N- terminal pro-BNP are currently under research as diagnostic marker of PDA. The primary mode of treatment for PDA is pharmacological closure using cyclo-oxygenase inhibitors with closure rate of 70-80%. Oral ibuprofen is emerging as a better alternative especially in Indian scenario where parenteral preparations of indomethacin are unavailable and side effects are comparatively lesser. Though pharmacological closure of PDA is an established treatment modality, there is still lack of evidence for long term benefits of such therapy as well as there is some evidence for the possible adverse effects like increased ROP and BPD rates, especially if treated prophylactically.The aim of this study is to investigate the effect of oral ibuprofen prophylaxis administrated on the first 24 hours of life and the following two days on hemodynamically significant patent ductus arterioses and its long term effects such as ROP and BPD.

DETAILED DESCRIPTION:
Patent ductus arterioses (PDA) is a major morbidity encountered in preterm neonates, especially in babies less than 28 weeks gestation or 1000g.Natural ductal closure is inversely related to gestational age and birth weight. The incidence ranges from 15% to 37% in newborn babies less than 1750 grams.The presence of PDA has significant effects on myocardial functions as well as systemic and pulmonary blood flow. Preterm newborns adapt, by increasing the left ventricular contractility, and thereby maintaining the effective systemic blood flow even when the left to right shunts equals 50% of the left ventricular output. This is mainly accomplished by an increase in stroke volume (SV)rather than heart rate.This increase in stroke volume is primarily due to reduction in afterload and simultaneous increase in left ventricular preload. An increasing number of biological substances like hormones, enzymes which are markers of cardiac stress, dysfunction or myocardial injury-collectively called biomarkers-are emerging as diagnostic and prognostic markers especially in the setting of heart failure or ischemic injury. The pharmacological basis for medical therapy is the use of non selective cyclo-oxygenase (COX) inhibitors, which inhibits prostaglandin synthesis and causes ductal constriction. The two most widely studied and used non selective COX inhibitors are indomethacin and ibuprofen. The future of pharmacological treatment of PDA could be with the use of nitric oxide inhibitors and prostaglandin receptor antagonists. Ibuprofen is an effective choice for the treatment of PDA in preterm infants as it has been demonstrated in previous several studies.Since there is a meta-analysis that claims there is no need for further studies about ibuprofen prophylaxis to treat PDA in low birth weight infants we aimed to evaluate the effect of ibuprofen prophylaxis in very extremely low birth weight infants. One such marker emerging in the diagnosis of hs-PDA is brain natriuretic peptide (BNP). Natriuretic peptides are hormones, produced either by atria (atrial natriuretic peptide-ANP) or by ventricles (BNP) in response to myocardial stress, secondary to dilatation, hypertrophy or increased wall tension.One of the aims of this study is to investigate the effect of oral prophylactic ibuprofen administration on BNP levels and renal functions.

ELIGIBILITY:
Inclusion Criteria:

* < 28 gestational week and/or < 1000 g birth weight preterm infants written parent consent

Exclusion Criteria:

* major congenital anomalies
* congenital heart diseases
* not having written parent consent

Ages: 23 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
the effect of oral ibuprofen to prevent hemodynamically significant PDA (hs-PDA) and from rescue therapy | in first week of life
  on the 3rd day of life all subjects will be examined by a experienced pediatric cardiologist and echocardiography will performed to investigate hs-PDA

SECONDARY OUTCOMES:
long term effects of oral ibuprofen prophylaxis in VELBW | corrected 36 weeks or until discharge
  long term effects such as ROP, BPD,IVH, duration of respiratory support and hospitalization are going to be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Zekai Tahir Burak Maternity Teaching Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Gokmen T, Erdeve O, Altug N, Oguz SS, Uras N, Dilmen U. Efficacy and safety of oral versus intravenous ibuprofen in very low birth weight preterm infants with patent ductus arteriosus. J Pediatr. 2011 Apr;158(4):549-554.e1. doi: 10.1016/j.jpeds.2010.10.008. Epub 2010 Nov 20. PMID 21094951
- [Background] Erdeve O, Gokmen T, Altug N, Dilmen U. Oral versus intravenous ibuprofen: which is better in closure of patent ductus arteriosus? Pediatrics. 2009 Apr;123(4):e763. doi: 10.1542/peds.2009-0003. No abstract available. PMID 19336363